CLINICAL TRIAL: NCT06657352
Title: Skin Efficacy Testing of Astrion Products
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Chia Nan University of Pharmacy ＆ Science (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: TSMHIRB22-111-A
Record Dates: First submitted 2024-10-23; First posted 2024-10-24 (Actual); Last update posted 2024-10-26 (Actual); Status verified 2024-10

CONDITIONS: Skin Pigment; Skin Red
MeSH Terms: conditions — Pigmentation Disorders; Erythema | interventions — Therapeutics

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (6):
- ACS Topical Treatment Group (Experimental): 25 participants, measured at Week 0, 2, 4.
  Interventions: Dietary Supplement: ACS Topical Treatment Group
- Topical Placebo Group (Placebo Comparator): 25 participants, measured at Week 0, 2, 4.
  Interventions: Dietary Supplement: Topical Placebo Group
- ACS Oral Treatment Group (Experimental): 25 participants, measured at Week 0, 2, 4, 8, 12.
  Interventions: Dietary Supplement: ACS Oral Treatment Group
- Oral Placebo Group (Placebo Comparator): 25 participants, measured at Week 0, 2, 4, 8, 12.
  Interventions: Dietary Supplement: Oral Placebo Group
- ACS Oral Treatment + ACS Topical Treatment Group (Experimental): 25 participants, measured at Week 0, 2, 4, 8, 12.
  Interventions: Dietary Supplement: Oral Treatment + Topical Treatment Group
- ACS Oral Treatment + Topical Placebo Group (Placebo Comparator): 25 participants, measured at Week 0, 2, 4, 8, 12.
  Interventions: Dietary Supplement: Oral Treatment + Topical Placebo Group

INTERVENTIONS:
Dietary Supplement: ACS Topical Treatment Group — The topical group applied the ACS cream to the face twice daily (morning and night) for 4 weeks.
  Arms: ACS Topical Treatment Group
Dietary Supplement: Topical Placebo Group — The topical group applied the cream (without ACS) to the face twice daily (morning and night) for 4 weeks.
  Arms: Topical Placebo Group
Dietary Supplement: Oral Treatment + Topical Treatment Group — The combination group used both the topical and oral ACS products for 12 weeks.
  Arms: ACS Oral Treatment + ACS Topical Treatment Group
Dietary Supplement: ACS Oral Treatment Group — The oral group ingested one ACS capsule twice daily after breakfast and dinner for 12 weeks.
  Arms: ACS Oral Treatment Group
Dietary Supplement: Oral Placebo Group — The oral group ingested one capsule (without ACS) twice daily after breakfast and dinner for 12 weeks.
  Arms: Oral Placebo Group
Dietary Supplement: Oral Treatment + Topical Placebo Group — The combination group used both the topical and oral products without ACS for 12 weeks.
  Arms: ACS Oral Treatment + Topical Placebo Group

SUMMARY:
This project aims to conduct safety and efficacy tests on the skin for the ingestion of Astrion Vitality Capsules, containing A. membranaceus and C. Asiatica roots, and the topical application of Astrion Vitality Cream. The goal is to develop health and skincare products that regulate physiological functions, promote overall wellness, and enhance skin beauty.

ELIGIBILITY:
Inclusion Criteria:

* Subjects aged ≥18 years.

Exclusion Criteria:

* Non-voluntary participants.
* Subjects diagnosed with skin diseases, cirrhosis, or chronic renal failure by a -physician.
* Individuals with known allergies to cosmetics, drugs, or food.
* Pregnant or breastfeeding women.
* Individuals taking medication for chronic diseases.
* Subjects who, within 12 weeks prior to the test, have undergone laser facial treatments, chemical peels, or experienced prolonged sun exposure (more than 3 hours of direct sunlight in a week).
* Students taught by the investigator.
* Individuals unwilling to allow the publication of photos of the experimental results.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 150 (Actual)
Dates: Start 2022-11-28 (Actual); Primary Completion 2023-09-30 (Actual); Study Completion 2023-09-30 (Actual)

PRIMARY OUTCOMES:
skin melanin | The topical group applied ACS cream to the face twice daily for 4 weeks. The oral group took one ACS capsule twice daily after meals for 12 weeks. The combination group followed both regimens for 12 weeks. A placebo group, identical in appearance but wit
  Skin elastometer (Soft Plus) was utilized to measure skin melanin. Units: arbitrary units
Skin brightness | The topical group applied ACS cream to the face twice daily for 4 weeks. The oral group took one ACS capsule twice daily after meals for 12 weeks. The combination group followed both regimens for 12 weeks. A placebo group, identical in appearance but wit
  Skin color difference analyzer (Chroma Meter MM500) was utilized to measure skin brightness
skin moisture | The topical group applied ACS cream to the face twice daily for 4 weeks. The oral group took one ACS capsule twice daily after meals for 12 weeks. The combination group followed both regimens for 12 weeks. A placebo group, identical in appearance but wit
  Skin moisture meter (Corneometer CM825) was utilized to measure skin moisture. Units: arbitrary units
skin elasticity | The topical group applied ACS cream to the face twice daily for 4 weeks. The oral group took one ACS capsule twice daily after meals for 12 weeks. The combination group followed both regimens for 12 weeks. A placebo group, identical in appearance but wit
  Skin elastometer (Soft Plus) was utilized to measure skin elasticity. Units: arbitrary units
collagen density content | The topical group applied ACS cream to the face twice daily for 4 weeks. The oral group took one ACS capsule twice daily after meals for 12 weeks. The combination group followed both regimens for 12 weeks. A placebo group, identical in appearance but wit
  Subcutaneous collagen scanner (DermaLab® Series SkinLab Combo) was utilized to measure skin collagen. Units: arbitrary units
skin surface topography | The topical group applied ACS cream to the face twice daily for 4 weeks. The oral group took one ACS capsule twice daily after meals for 12 weeks. The combination group followed both regimens for 12 weeks. A placebo group, identical in appearance but wit
  VISIA Micro-Analysis Skin Image Analyzer was utilized to measure skin texture. Units: arbitrary units

CONTACTS AND LOCATIONS:
Locations (1):
- Chia Nan University of Pharmacy ＆ Science, Tainan, Taiwan

IPD SHARING:
Plan to Share IPD: No